CLINICAL TRIAL: NCT03409666
Title: Randomized Controlled Study Comparing the Taperloc Complete Versus the Taperloc Complete Microplasty.
Brief Title: Randomized Controlled RSA Study Comparing the Taperloc Complete Versus the Taperloc Complete Microplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO.CR.GH60
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Hip Osteoarthritis; Noninflammatory Degenerative Joint Disease; Avascular Necrosis; Correction of Functional Deformity; Rheumatoid Arthritis
Keywords: Total Hip Arthroplasty; Medical Device; Performance; Safety; Hip prosthesis; Roentgen Stereophotogrammetric Analysis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteonecrosis; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: 1:1 assignment of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Taperloc Complete Microplasty stem (Experimental): Subjects in need of a total hip artthroplasty who received the Taperloc Complete Microplasty stem.
  Interventions: Device: Taperloc Complete Microplasty stem
- Taperloc Complete Reduced Distal stem (Active Comparator): Subjects in need of a total hip arthroplasty who received the Taperloc Complete Reduced Distal stem.
  Interventions: Device: Taperloc Complete Reduced Distal stem

INTERVENTIONS:
Device: Taperloc Complete Microplasty stem — Total hip replacement with Taperloc Complete Microplasty stem and G7 acetabular shell with E1 liner
  Other Names: Total hip arthroplasty
  Arms: Taperloc Complete Microplasty stem
Device: Taperloc Complete Reduced Distal stem — Total hip replacement with Taperloc Complete Reduced Distal stem and G7 acetabular shell with E1 liner
  Other Names: Total hip arthroplasty
  Arms: Taperloc Complete Reduced Distal stem

SUMMARY:
This is a single center, prospective, randomized controlled study. The primary objective of this study is to measure migration over two years with RSA. Patients will be randomized in two arms, receiving a Taperloc Complete Reduced Distal or a Taperloc Complete Microplasty hip stem.

DETAILED DESCRIPTION:
A total of 50 patients will be enrolled into the study, randomized 1:1. All patients will receive a G7 limited hole acetabular cup with E1 liner.

All potential study subjects will be required to participate in the Informed Consent process.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis, avascular necrosis and rheumatoid arthritis.
* Correction of functional deformity.
* Male or female

  -≥ 18 and ≤ 70 years of age
* Subjects willing to return for follow-up evaluations.
* Subjects able to read and understand Dutch language.

Exclusion Criteria:

* active Infection (or within 6 weeks after infection)
* Sepsis
* Osteomyelitis
* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* diagnosed Osteoporosis or Osteomalacia
* Metabolic disorders which may impair bone formation
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy or neuromuscular disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, BSc, Study Director — Zimmer Biomet
Locations (1):
- Bravis, Roosendaal, Netherlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Started | 25 | 25
Completed | 25 | 21
Not Completed | 0 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Population: These numbers represent the subjects who received either the Taperloc Complete Microplasty stem or the Taperloc Complete Reduced Distal stem.
  25 patients were enrolled in the TCM group, and 25 in the TCRD group. In the TCM group, 1 patient was withdrawn before surgery. In the TCRD group, 3 received a different device, and 1 the TCM. For clarity, we decided to report based on the actual implantation (i.e. 25 TCM and 21 TCRD).
Groups:
- Total: Total of all reporting groups
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem | Total
Number analyzed (Participants) | 25 | 21 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: These numbers represent the subjects who received either the Taperloc Complete Microplasty stem or the Taperloc Complete Reduced Distal stem.
  25 patients were enrolled in the TCM group, and 25 in the TCRD group. In the TCM group, 1 patient was withdrawn before surgery. In the TCRD group, 3 received a different device, and 1 the TCM. For clarity, we decided to report based on the actual implantation (i.e. 25 TCM and 21 TCRD).
  years | 63.6 (6.3) | 63.9 (6.5) | 63.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: These numbers represent the subjects who received either the Taperloc Complete Microplasty stem or the Taperloc Complete Reduced Distal stem.
  25 patients were enrolled in the TCM group, and 25 in the TCRD group. In the TCM group, 1 patient was withdrawn before surgery. In the TCRD group, 3 received a different device, and 1 the TCM. For clarity, we decided to report based on the actual implantation (i.e. 25 TCM and 21 TCRD).
  Participants
    Female | 20 | 15 | 35
    Male | 5 | 6 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Stability Over a Period of Two Year Measured by Migration With Röntgen Stereophotogrammetric Analysis (RSA)
Description: Migration and rotation in three directions represented by Maximum Total Point Motion (MTMP)
Time Frame: 2 years postoperatively
Population: RSA data from 35 patients (20 Taperloc Complete Reduced Distal & 15 Taperloc Complete Microplasty) is available for the comparison of migration between the investigated stems.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Number analyzed (Participants) | 15 | 20
mm | 3.15 (2.40) | 3.90 (4.17)

2. Secondary Outcome: Difference in Surgical Positioning Between Taperloc Complete Reduced Distal and Taperloc Complete Microplasty
Description: Assessed by difference in the prevalence of stem malalignment, incorrect sizing and subsidence based on radiographic evaluation.
Time Frame: 2 years postoperatively
Measure: Number; unit: participants
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Number analyzed (Participants) | 25 | 21
participants
  Stem malalignment | 0 | 0
  Incorrect sizing | 0 | 0
  Subsidence | 2 | 6

3. Secondary Outcome: Early Survival Assessed by Counting the Number of Implant Revisions
Description: Assessed by counting the number of implant revisions
Time Frame: Immediate post-operatively, 6 weeks, 1 year and 2 years postoperatively
Measure: Number; unit: implant revisions
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Number analyzed (Participants) | 25 | 21
implant revisions | 0 | 0

4. Secondary Outcome: Clinical Performance Measured by Clinician Based Outcome Sore Harris Hip Score (HHS)
Description: Harris Hip Score (HHS), a score to measure health and satisfaction after a hip prosthesis.
  The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points)
Time Frame: pre-operatively (within 3 months of surgery), 6 weeks, 1 year and 2 years postoperatively
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Number analyzed (Participants) | 25 | 21
scores on a scale
  pre-op | 63.9 (7.7) | 65.1 (13.9)
  6 week | 79.9 (11.4) | 82.4 (8.8)
  1 year | 96.7 (4.6) | 95.7 (5.9)
  2 year | 98.3 (3.1) | 97.6 (4.9)

5. Secondary Outcome: Clinical Performance Measured by Clinician Based Outcome Radiological Evaluation
Description: Assess radiographs for signs of stress shielding, radiolucency and stem alignment.
Time Frame: 6 weeks, 1 year and 2 years postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Number analyzed (Participants) | 25 | 21
Participants
  Stress shielding | 0 | 0
  Radiolucency | 0 | 0
  stem alignment (between <5 valgus and <5 varus) | 25 | 21

6. Secondary Outcome: Clinical Performance Measured by Patient Based Outcome Using Hip Disability and Osteoarthritis Outcome Score (HOOS)
Description: The outcomes of the subcategories are scored on a 0 to 100 scale, with 100 indicating no symptoms.
Time Frame: 2 years postoperatively
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Number analyzed (Participants) | 25 | 21
scores on a scale
  Pain | 94.2 (10.5) | 92 (9.2)
  Symptoms | 89.8 (12) | 85.5 (13.3)
  Activity limitations daily living | 92.7 (11.4) | 90.8 (10.1)
  Sport/Recreation | 80.7 (24.1) | 79.6 (20.2)
  Quality of life | 89.7 (16.8) | 84.4 (17)

7. Secondary Outcome: Clinical Performance Measured by Patient Based Outcome EQ5D
Description: Each question in the EQ5D assessment can be answered in three ways, indicating no, moderate or extreme problems. Index scores are created with a weight for each dimension, ranging from 0 (health state equivalent to death) to 1 (perfect health). The EQ5D also includes a question about health status, ranging from 0 (worst health) to 100 (best health).
Time Frame: 2 years postoperatively
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Number analyzed (Participants) | 24 | 20
score on a scale
  EQ-5D | 0.9 (0.1) | 0.9 (0.1)
  Health status | 81.0 (12.3) | 81.0 (15.6)

8. Secondary Outcome: Clinical Performance Measured by Patient Based Outcome Using Oxford Hip Score (OHS)
Description: The OHS assesses pain (6 items) and function (6 items) of the hip in relation to daily activities such as walking, dressing, sleeping, etc. The scoring is the following: 0-4 (worst to best) with overall scores ranging from 0-48 where 48 represents the best score.
Time Frame: pre-operatively(within 3 months of surgery), 6 weeks, 1 year and 2 years postoperatively
Population: Number of analyzed patients differs between the time points due to missing values
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Number analyzed (Participants) | 25 | 21
scores on a scale
  pre-op: number analyzed (Participants) | 25 | 20
  pre-op | 26.1 (7.6) | 25.6 (8.5)
  6 week: number analyzed (Participants) | 24 | 21
  6 week | 38.3 (6.7) | 37.5 (4.8)
  1 year: number analyzed (Participants) | 25 | 20
  1 year | 44.6 (3.4) | 43.1 (4.1)
  2 year: number analyzed (Participants) | 24 | 20
  2 year | 45.7 (3.8) | 44.9 (3.6)

9. Secondary Outcome: Clinical Performance Measured by Patient Based Outcome Forgotten Joint Score (FJS)
Description: The Forgotten Joint Score (FJS) is a questionnaire, which focuses on the awareness of having a joint prosthesis.
  The rationale of this questionnaire is that the ultimate goal in joint arthroplasty resulting in the greatest possible patient satisfaction is the ability to forget the artificial joint. The outcome is scored on a 0 to 100 scale, with a total score of 0 indicating the highest level of awareness of having a joint prosthesis.
Time Frame: 6 weeks, 1 year and 2 years postoperatively
Population: Number of analyzed patients differs between the time points due to missing values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
Number analyzed (Participants) | 25 | 21
score on a scale
  6 week | 47.8 (30) | 43.2 (26.1)
  1 year: number analyzed (Participants) | 25 | 20
  1 year | 69.9 (29.2) | 61.7 (29.6)
  2 year: number analyzed (Participants) | 23 | 19
  2 year | 72.3 (30.5) | 80.3 (26.5)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Taperloc Complete Microplasty Stem | Taperloc Complete Reduced Distal Stem
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/25 | 0/21
Other Adverse Events (participants affected / at risk) | 2/25 | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Taperloc Complete Microplasty Stem (N=25) | Taperloc Complete Reduced Distal Stem (N=21)
Fever (General disorders) | 1 | 0
hypotension (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Taperloc Complete Microplasty Stem (N=25) | Taperloc Complete Reduced Distal Stem (N=21)
Stem Subsidence (Musculoskeletal and connective tissue disorders) | 2 | 6
Periarticular Ossification (Musculoskeletal and connective tissue disorders) | 0 | 1 — Other hip related radiographic finding
Pedestal Sign (Musculoskeletal and connective tissue disorders) | 0 | 2 — Other hip related radiographic finding

LIMITATIONS AND CAVEATS:
A limitation of the study was that 14 patients had to be excluded for RSA analysis due to insufficient bone markers or not meeting other criteria to perform an accurate RSA migration calculation. However, as Valstar et al. (2005) stated that at least 15-25 patients are needed per group, we believe that the results of this study are still valuable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03409666/Prot_SAP_000.pdf